CLINICAL TRIAL: NCT06226025
Title: Correcting Circadian Rhythms to Breakthrough in Bipolar Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leslie Swanson (Other)
Collaborators: University of Michigan (Other); Natrol (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Leslie Swanson, Associate Professor of Psychiatry, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00235778; 1R21MH132901-01A1 (NIH)
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Bipolar Disorder; Delayed Sleep-Wake Phase Disorder
Keywords: Correcting Circadian Rhythms; Melatonin; Placebo; Dim light melatonin onset
MeSH Terms: conditions — Bipolar Disorder; Sleep Disorders, Circadian Rhythm | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Participants that meet eligibility for the randomized trial are randomized using minimization in a 1:1 ratio to low-dose afternoon melatonin plus a behavioral sleep intervention (MEL) or placebo tablet plus behavioral sleep placebo (CTL)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): Oral medication will be taken for 28 days on the afternoon or evening of the participants first intervention session and continue daily for the remainder of the treatment period.
  Interventions: Drug: Melatonin; Behavioral: Behavioral sleep intervention
- Placebo (Placebo Comparator): Oral medication will be taken for 28 days on the afternoon or evening of the participants first intervention session and continue daily for the remainder of the treatment period.
  Interventions: Other: Placebo; Behavioral: Behavioral sleep control

INTERVENTIONS:
Drug: Melatonin — Participants randomized to this intervention will take 1 oral pill (0.5 milligrams (mg)) daily. They will attend 4 weekly behavioral sleep intervention sessions with a therapist. In addition, participants will complete questionnaires (MyDataHelp app), monitor sleep, collect saliva samples, and wear the Fitbit Device.
  Arms: Melatonin
Other: Placebo — Participants randomized to this intervention will take 1 oral placebo pill daily. They will attend 4 weekly behavioral sleep control sessions with a therapist. In addition, participants will complete questionnaires (MyDataHelp app), monitor sleep, collect saliva samples, and wear the Fitbit Device.
  Arms: Placebo
Behavioral: Behavioral sleep intervention — An active intervention that is typically paired with melatonin to maximize treatment effects.
  Arms: Melatonin
Behavioral: Behavioral sleep control — A behavioral placebo (which does not improve sleep in delayed sleep-wake phase disorder) to control for social/interpersonal effects of behavioral sleep intervention sessions.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether a dietary supplement (low-dose melatonin) commonly used to treat night owls, administered in conjunction with a behavioral sleep intervention, will help to shift the brain clock earlier and improve mood and sleep in bipolar disorder. Eligible participants will be randomized to receive melatonin plus a behavioral sleep intervention or placebo plus a behavioral sleep placebo.

The hypotheses for this study include:

* Melatonin plus behavioral sleep intervention (compared to placebo plus behavioral sleep placebo) will produce a greater advance of dim light melatonin onset (DLMO), between pre- and post-treatment.
* Melatonin (compared to placebo) will produce a greater reduction in Patient Health Questionnaire-9 score between pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Meet The Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria for bipolar disorder (BD) I or II
* Evening chronotype per the Morningness-Eveningness Questionnaire (MEQ) defined by a score of <42
* At least mild depressive symptoms on the Patient Health Questionnaire (PHQ)-9 defined by a score ≥5
* Psychotropic medications at stable dose for past month
* Able to download the MyDataHelps mobile application (app), and open app on participants' own phone
* Willing to abstain from alcohol for the duration of the intervention phase
* Female participants of childbearing potential (i.e., patients are not permanently sterilized (hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) or postmenopausal (12 months with no menses without an alternative medical cause) by report) must agree to use a reliable method of contraception from the screening visit until 4 weeks after the study has completed.

Exclusion Criteria:

* Current diagnosis of, or high risk for, a sleep disorder other than DSPD per interview and medical record review (when available) including:

  * Insomnia per DSM-5
  * Sleep-disordered breathing per Snoring, tiredness, observed apnea, blood pressure, body mass index, age, neck circumference, and gender (STOP-BANG)
  * Restless leg syndrome per sleep interview
  * Narcolepsy
  * Suspicion of vasomotor symptoms impacting sleep per interview for women that may be perimenopausal or postmenopausal.
* Risk of current mania (per Young Mania Rating Scale (YMRS) score > 19).
* Suicidal or at high risk for suicide per Columbia Suicide Severity Rating Scale (C-SSRS) guidelines (i.e., presence of any suicidal behavior-suicide attempt, interrupted attempt, abort attempt, or preparatory behavior-in the past 3 months; and/or current active suicidal ideation with any intent), or as determined by the principal investigators.
* Presence of cardiac implantable electronic device, such as defibrillator or pacemaker.
* Presence of chronic psychiatric conditions which may directly influence sleep per interview and medical record review (when available), including:

  * Current illicit drug use per the Drug Use Disorders Identification Test (DUDIT) defined by a score of ≥ 25
  * Current alcohol or drug abuse per the Alcohol Use Disorder Identification Test (AUDIT) defined by a score of ≥ 16 and DUDIT
  * Currently experiencing psychosis
* Presence of unstable chronic medical condition which may directly influence sleep:

  * Chronic pain
  * Thyroid conditions
* Current or history of medical conditions which may be affected by melatonin per self-report and medical record review (when available), such as:

  * Hypertension or hypotension
  * Diabetes Type 1 or Type 2
  * Clotting/bleeding disorders
  * Epilepsy/seizures
  * Autoimmune disorders
  * Conditions requiring immunosuppressive management such as transplant
* Per self-report or medical record review (when available), current use of medications which may have interactions with melatonin (see protocol for more details).
* Current use of medications that may interfere with the measurement of melatonin (non-steroidal anti-inflammatory drugs if used daily, and beta-blockers), per self-report and medical record review (when available).
* Self-report use of melatonin in the past month.
* Hypersensitivity to melatonin or any other component of the melatonin or placebo product.
* Pregnancy (as determined by dipstick urinary pregnancy test at screening for women of child-bearing potential) or self-report of breastfeeding and/or plan to become pregnant in the next 3 months.
* Self-report of routine night shift work.
* Self-report of past month travel or planned travel during the study across more than one time zone.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in time of Dim Light Melatonin Onset (DLMO) baseline (pre-treatment) to 4 weeks (post-treatment) | 4 weeks (after treatment period)
  Onset of melatonin in dim light conditions as measured in saliva (also called DLMO). Time of DLMO is measured in clock time and change in time of DLMO is measured in hours. The change score is calculated as time at 4 weeks minus baseline time. Thus, positive scores indicate a shift towards a later onset of melatonin and negative scores indicate a shift towards an earlier onset of melatonin.

SECONDARY OUTCOMES:
Change in the Patient Health Questionnaire-9 (PHQ-9) | Baseline, 4 weeks (after treatment period)
  The PHQ-9 is a 9-item self-report scale to screen for symptoms of depression. Items are rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 27, where higher scores indicate more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Swanson, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Additional data collected as part of the study's fundings requirements per the National Institute of Mental Health to be shared to the National Institute of Mental Health Data Archive include the Generalized Anxiety-Disorder 7 item scale; World Health Organization Disability Assessment Schedule 2.0 scale, and the DSM-5 cross cutting assessment. Under the current protocol these data are to be collected to fulfill the National Institute of Mental Health funding requirements but are not included as endpoints or in our analytic plan.
Supporting Information: Study Protocol, SAP, ICF